CLINICAL TRIAL: NCT00595296
Title: GeneSearch™ Breast Lymph Node (BLN) Assay Post Approval Study
Status: Terminated | Type: Observational
Why Stopped: GeneSearch™ BLN Assay has been voluntarily withdrawn from the US market.
Sponsor: Janssen Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: GeneSearch BLN Assay PPC Study; BLN-US-2007.00
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: BreastCancer; Sentinel Lymph Nodes; Metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Biological Assay

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of the lymph node tissue homogenate and RNA extract are collected if the subject gives permission via the informed consent form.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All eligible patients.
  Interventions: Device: GeneSearch™ Breast Lymph Node (BLN) Assay

INTERVENTIONS:
Device: GeneSearch™ Breast Lymph Node (BLN) Assay — The GeneSearch™ BLN Assay is a real time Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) assay that detects the presence of breast tumor cell metastasis in lymph nodes through the detection of gene expression markers present in breast tissue, but not in nodal tissue (cell type specific messenger RNA).
  Other Names: BLN Assay; GeneSearch™ BLN Assay

SUMMARY:
This post-approval study is designed to determine the performance of the FDA-approved GeneSearch™ BLN Assay when compared to the site's standard of care permanent section histological evaluation, and when compared to more extensive histological evaluation when the assay is being used by clinicians to make surgical decisions on complete axillary dissections (ALND).

DETAILED DESCRIPTION:
The primary objective of this clinical study is to gather data to estimate the positive predictive concordance (PPC) between the GeneSearch™ BLN Assay and histology as routinely practiced, i.e., routine H&E histology of sentinel lymph node(s) (SLN) and, when available, routine histology of non-sentinel axillary lymph nodes (ALN). This study will provide information on the assay that will augment the performance data gained in pre-market validation studies. In addition, with the assay being used for ALND decision-making, the metastatic status of the non-sentinel axillary nodes can be taken into account in the performance measures, i.e., if the patient's sentinel or non-sentinel nodes are histologically positive, the patient will be considered positive for the primary comparison to the assay results.

ELIGIBILITY:
Inclusion Criteria:

* Pre-operatively established diagnosis of invasive carcinoma of the breast
* Scheduled for axillary sentinel lymph node dissection as per standard of care at the clinical site for newly diagnosed breast cancer patients
* Patients for whom the GeneSearch™ BLN Assay will be used intra-operatively to make a decision for an axillary lymph node dissection
* 18 years of age or older
* Female or male
* Willing and able to give informed consent to participate in the study

Exclusion Criteria:

* Previous diagnosis of lymphoma
* Subjects participating in other research studies that would interfere with their full participation in this study
* Patients and/or conditions with 'interfering substances' as listed in the IFU.
* Patients who have had any pre-operative treatment for breast cancer including neoadjuvant and/or hormonal intervention such as aromatase inhibitors or tamoxifen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have been diagnosed with carcinoma of the breast and be a candidate for lymph node surgery as per each site's standard of care. The patients may be female or male, at least 18 years old, and must meet study inclusion criteria described later in this protocol. Patients receiving pre-operative therapy for breast cancer, such as neoadjuvant therapy and/or hormonal intervention are not eligible to participate in this study.
Sampling Method: Probability Sample
Enrollment: 461 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To estimate the positive predictive concordance (PPC) between the GeneSearch™ BLN Assay and histology as routinely practiced. | 1 week

SECONDARY OUTCOMES:
To estimate the positive predictive value (PPV) of the GeneSearch™ BLN Assay as measured against histology that is as accurate as possible in assessing whether a SLN is truly positive. | 1 week
To gather data on size of metastases (micrometastases versus macrometastases) identified by histology to examine the assay performance for various levels of metastases. | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Scott U Adams, MS, Study Director — Ortho-Clinical Diagnostics, Inc.
Locations (6):
- United States (6):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - St. Anthony's Hospital, St. Petersburg, Florida
  - Georgia Esoteric and Molecular Labs, LLC, Augusta, Georgia
  - Woman's Hospital, Flowood, Mississippi

REFERENCES:
- [Background] Blumencranz P, Whitworth PW, Deck K, Rosenberg A, Reintgen D, Beitsch P, Chagpar A, Julian T, Saha S, Mamounas E, Giuliano A, Simmons R. Scientific Impact Recognition Award. Sentinel node staging for breast cancer: intraoperative molecular pathology overcomes conventional histologic sampling errors. Am J Surg. 2007 Oct;194(4):426-32. doi: 10.1016/j.amjsurg.2007.07.008. PMID 17826050
- [Background] Julian TB, Blumencranz P, Deck K, Whitworth P, Berry DA, Berry SM, Rosenberg A, Chagpar AB, Reintgen D, Beitsch P, Simmons R, Saha S, Mamounas EP, Giuliano A. Novel intraoperative molecular test for sentinel lymph node metastases in patients with early-stage breast cancer. J Clin Oncol. 2008 Jul 10;26(20):3338-45. doi: 10.1200/JCO.2007.14.0665. PMID 18612150
- [Background] Veys I, Majjaj S, Salgado R, Noterman D, Schobbens JC, Manouach F, Bourgeois P, Nogaret JM, Larsimont D, Durbecq V. Evaluation of the histological size of the sentinel lymph node metastases using RT-PCR assay: a rapid tool to estimate the risk of non-sentinel lymph node invasion in patients with breast cancer. Breast Cancer Res Treat. 2010 Dec;124(3):599-605. doi: 10.1007/s10549-009-0555-2. Epub 2009 Sep 25. PMID 19779817